CLINICAL TRIAL: NCT05318963
Title: A Phase I, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LCAR-AIO, a Triple-targeted Cell Preparation Targeting CD19/CD20/CD22, in Patients With Relapsed/Refractory B-cell Lymphoma
Brief Title: Targeting CD19/CD20/CD22 Triple-targeted Cell in Patients With Relapsed/Refractory B-cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The collaborators decided to terminate this study.
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021066
Record Dates: First submitted 2022-03-15; First posted 2022-04-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-AIO cells product (Experimental): Each subject will be given a single-dose LCAR-AIO cells infusion at each dose level.
  Interventions: Biological: LCAR-AIO cells product

INTERVENTIONS:
Biological: LCAR-AIO cells product — before treatment with LCAR-AIO cells, subjects will receive a conditioning regimen (IV infusion of cyclophosphamide 300 mg/m^2 and fludarabine 30mg/m^2 once daily (QD) for 3 days.

SUMMARY:
A phase I, open-label clinical study to evaluate the safety, tolerability, and efficacy of LCAR-AIO, a triple-targeted cell preparation targeting CD19/CD20/CD22, in patients with relapsed/refractory B-cell lymphoma.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation/dose extension study to assess the safety, tolerability, and efficacy of LCAR-AIO in the patient ≥ 18 years of age with relapsed or refractory B cell lymphoma. Subjects who meet the eligibility criteria will receive a single dose of LCAR-AIO injection. The study will include the following sequential phases: screening, pre-treatment (cell product preparation; lymphodepleting chemotherapy), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have fully understood the possible risks and benefits of participating in this study, are willing to follow and able to complete all trial procedures, and have signed informed consent.
2. Aged 18-75 years (inclusive).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed B-cell lymphoma that expresses at least one of CD19/CD20/CD22.
5. At least one measurable tumor lesion determined according to Lugano 2014 criteria.
6. Response to prior therapy is consistent with one of the following:

   1. Primary refractory: it means that the best response to first-line therapy (at least 2 cycles) is PD, or best response to first-line therapy (at least 4 cycles) is SD but the duration is less than 6 months, which is considered to be PD;
   2. Relapsed or refractory after 2 or more lines of therapy. Refractory is defined that best respond to the most recent treatment regimen (at least 2 cycles) is PD, or best response to the most recent treatment regimen (at least 4 cycles) is SD but the duration is less than 6 months, which is considered to be PD;
   3. Progression or relapse within 12 months after hematopoietic stem cell transplantation; if salvage therapy is applied after transplantation, the patient must be unresponsive or relapsed to the last line of therapy;
7. Life expectancy≥ 3 months
8. Clinical laboratory values meet screening visit criteria
9. Adequate organ function;

Exclusion Criteria:

Subject eligible for this study must not meet any of the following criteria:

1. Prior antitumor therapy with insufficient washout period ;
2. Patients who received dual-targeted CAR-T cell therapy (including but not limited to sequential infusion) at any time in the past, or who received CAR-T cell therapy of cameloid origin;
3. With acute or chronic graft-versus-host disease (GvHD);
4. Patients who are positive for any index of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), or human immunodeficiency virus antibody (HIV- Ab).
5. Known life-threatening allergies, hypersensitivity, or intolerance to LCAR-AIO CAR-T cell or its excipients, including DMSO (refer to Investigator's Brochure).
6. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and type of TEAEs (Treatment-emergent Adverse Events) | Minimum 2 years after LCAR-AIO infusion (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Pharmacokinetics in peripheral blood | Minimum 2 years after LCAR-AIO infusion (Day 1)
  CAR positive T cells and CAR transgene levels in peripheral blood after LCAR-AIO infusion.
Pharmacokinetics in bone marrow | Minimum 2 years after LCAR-AIO infusion (Day 1)
  CAR positive T cells and CAR transgene levels in bone marrow after LCAR-AIO infusion.
The recommended Phase II dose (RP2D) for this cell therapy | 30 days after LCAR-AIO infusion
  RP2D established through ATD+BOIN design and the DLTs occurring following CAR T-cell infusion

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, minimum 2 years after LCAR-AIO infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LCAR-AIO cell infusion
Progression-free survival (PFS) | Through study completion, minimum 2 years after LCAR-AIO infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LCAR-AIO to the first documented disease progression (according to Lugano 2014) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Through study completion, minimum 2 years after LCAR-AIO infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-AIO to death of the subject
Time to Response (TTR) | Through study completion, minimum 2 years after LCAR-AIO infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LCAR-AIO to the date of the first response evaluation of the subject who has met all criteria for CR or PR.
Duration of Response (DoR) | Through study completion, minimum 2 years after LCAR-AIO infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or PR) to the first documented relapse evidence of the responders
Immunogenicity assessment of LCAR-AIO cells | Through study completion, minimum 2 years after LCAR-AIO infusion (Day 1)
  The incidence of Anti-LCAR-AIO antibody in patients who received LCAR-AIO cells infusion

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gobroad Boren Hospital, Beijing, Beijing Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No